CLINICAL TRIAL: NCT00701922
Title: Season Surveillance Study of Viral Infections in Lung Transplant Recipients
Brief Title: Surveillance Study of Viral Infections Following Lung Transplantation
Status: Completed | Type: Observational
Sponsor: Hannover Medical School (Other)
Collaborators: Department of Pulmonology (Unknown); Department of Virology (Ambiguous)
Responsible Party: Hannover Medical School, Hannover Medical School
Other Study IDs: 4015
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Last update posted 2011-10-28 (Estimated); Status verified 2008-12

CONDITIONS: Lung Transplantation; Bronchiolitis Obliterans; Epstein-Barr Virus Infections; Paramyxoviridae Infections
Keywords: lung transplantation; Bronchiolitis Obliterans; Epstein-Barr Virus Infections; Paramyxoviridae Infections; Herpesviridae
MeSH Terms: conditions — Bronchiolitis Obliterans; Epstein-Barr Virus Infections; Paramyxoviridae Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasopharyngeal and oropharyngeal swabs
  bronchoalveolar lavage
  blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The present study was conducted to study the impact community acquired respiratory virus (CARV) infections in an outpatient setting on graft function of lung transplant recipients. The study was aimed to identify risk factors for CARV infections.

The study was further intended to investigate an association of Epstein-Barr virus (EBV), cytomegalovirus (CMV) and human adenovirus (HAdV) with the development of BOS and to identify risk factors for virus detection in blood.

DETAILED DESCRIPTION:
Informed consent was obtained from the LTx recipients and the study was approved of by the institutional review board of Hannover medical school.

LTx recipients are screened for CARV infections during the cold season (end October until end April) in a single-centre outpatient clinic. Symptoms of upper (URTI) and lower respiratory tract infections (URTI) are recorded by questionnaires and findings.

Nasopharyngeal and oropharyngeal swabs (NOS) were performed to detect RV-antigens by immunofluorescence testing (IFT) of respiratory-syncytial virus (RSV), adenovirus, parainfluenza (PIV), influenza and cultures for CARV are performed. BAL was performed when clinically indicated and processed by IFT. Multiplex-PCR to detect 14 CARV are processed in symptomatic patients.

In addition blood samples are monitored at each contact to investigate an association of Epstein-Barr virus (EBV), cytomegalovirus (CMV) and human adenovirus (HAdV) with the development of BOS and to identify risk factors for virus detection in blood.

ELIGIBILITY:
Inclusion Criteria:

* adults 18-70 years
* lung transplantation (including single, double, combination and re-do transplants)

Exclusion Criteria:

* refused consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: lung transplant recipients in in a single-centre outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 388 (Actual)
Dates: Start 2005-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Incidence of bronchiolitis obliterans syndrome | 1 year

SECONDARY OUTCOMES:
Incidence of acute rejection | 1 year
Incidence of hospitalisation | 1 year
Incidence of graft loss (death or re-do-transplantation) | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Jens T Gottlieb, MD, Principal Investigator — Dpt. Pulmonary Medicine; Ilka Engelmann, MD, Principal Investigator — Dpt. Virology, MHH
Locations (1):
- Hannover Medical School, Hanover, Germany

REFERENCES:
- [Background] Khalifah AP, Hachem RR, Chakinala MM, Schechtman KB, Patterson GA, Schuster DP, Mohanakumar T, Trulock EP, Walter MJ. Respiratory viral infections are a distinct risk for bronchiolitis obliterans syndrome and death. Am J Respir Crit Care Med. 2004 Jul 15;170(2):181-7. doi: 10.1164/rccm.200310-1359OC. Epub 2004 May 6. PMID 15130908
- [Background] Kumar D, Erdman D, Keshavjee S, Peret T, Tellier R, Hadjiliadis D, Johnson G, Ayers M, Siegal D, Humar A. Clinical impact of community-acquired respiratory viruses on bronchiolitis obliterans after lung transplant. Am J Transplant. 2005 Aug;5(8):2031-6. doi: 10.1111/j.1600-6143.2005.00971.x. PMID 15996256
- [Background] Milstone AP, Brumble LM, Barnes J, Estes W, Loyd JE, Pierson RN 3rd, Dummer S. A single-season prospective study of respiratory viral infections in lung transplant recipients. Eur Respir J. 2006 Jul;28(1):131-7. doi: 10.1183/09031936.06.00105505. Epub 2006 Mar 1. PMID 16510454
- [Derived] Engelmann I, Welte T, Fuhner T, Simon AR, Mattner F, Hoy L, Schulz TF, Gottlieb J. Detection of Epstein-Barr virus DNA in peripheral blood is associated with the development of bronchiolitis obliterans syndrome after lung transplantation. J Clin Virol. 2009 May;45(1):47-53. doi: 10.1016/j.jcv.2009.02.005. Epub 2009 Mar 20. PMID 19303808